CLINICAL TRIAL: NCT01923649
Title: SOMATULINE Autogel 90 mg IN DUMPING SYNDROME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S50966; 2008-000643-34 (EudraCT Number)
Record Dates: First submitted 2013-07-19; First posted 2013-08-15 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2017-07

CONDITIONS: Dumping Syndrome
Keywords: postoperative dumping; somatostatin analogues; somatulin; lanreotide; dumping syndrome
MeSH Terms: conditions — Dumping Syndrome | interventions — lanreotide; Delayed-Action Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lanreotide slow release 90 mg (Experimental): Patients receive lanreatide slow release (Somatuline autogel) 90 mg every four weeks via a deep subcutaneous injection, three times. After a wash out period of 4 weeks they receive a similar placebo every for weeks, three times.
  Interventions: Drug: Lanreotide 90 mg slow release formulation
- Placebo (Placebo Comparator): Patients receive a deep subcutanous injection of placebo every four weeks, three times. After a wash out of three weeks, they will receive somatuline 90 mh via a deep subcutanous injection every four weeks, three times.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanreotide 90 mg slow release formulation — Lanreotide 90 mg slow release formulation is injected deep subcutaneously, every 4 weeks, three times and compared to placebo
  Other Names: Somatulin autogel
  Arms: Lanreotide slow release 90 mg
Drug: Placebo — Placebo for somatuline slow release 90 mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if Somatuline autogel 90 mg is effective in the treatment of dumping syndrome.

DETAILED DESCRIPTION:
Dumping syndrome has characteristic alimentary and systemic manifestations. It is one of the most common postprandial syndromes observed after extensive gastric surgery. Dumping syndrome can be separated into an early and late phase depending on the occurrence of symptoms in relation to the time elapsed after a meal. The early phase occurs because of rapid delivery of large amounts of osmotic active solids and liquids into the duodenum. The late phase is caused by a rapid increase of the glycemia and insuline causing hypoglycemia when the nutrients are not available any more. Dumping syndrome is the direct result of alterations in the storage function of the stomach and/or the pyloric emptying mechanism.

Incidence and severity of symptoms in dumping syndrome are related directly to the extent of gastric surgery. An estimated 25-50% of all patients who have undergone gastric surgery have some symptoms of dumping. Only 1-5% are reported to have severe disabling symptoms. Incidence of significant dumping has been reported to be 6-14% in patients after truncal vagotomy and drainage and from 14-20% in patients after partial gastrectomy. Incidence of dumping syndrome after proximal gastric vagotomy without any drainage procedure is less than 2%. In the pediatric population, dumping syndrome is described in children who have undergone Nissen fundoplication.

Several treatments can be proposed to a patient with dumping. Initially a diet of several small meals with a low concentration of mono-and disaccharides is prescribed and the patient is asked to avoid liquids during a meal. Several medical treatments can be utilized as guar gum, to increase the viscosity and reduce gastric emptying; pectine, to avoid a late hypoglycemia; acarbose, to block the digestion of saccharides. Some of them have only a partial effect or important side effects.

Surgical interventions like an interposition of an antiperistaltic jejunal segment will reduce the intestinal motility or a Roux-en-Y construction can be created. These surgical interventions are sometimes necessary but remain quite invasive and not always useful.

Somatostatin analogues have been used with success in patients with dumping syndrome. They exert a strong inhibitory effect on the release of insulin and several gut-derived hormones. The effectiveness of analogues in controlling the symptoms of both early and late dumping has been demonstrated in several randomized control trials. Somatostatin analogues interfere with the pathophysiology of a dumping syndrome in several ways. Somatostatin analogues reduce the secretion of insulin and prevents the occurrence of a late hypoglycaemia; decrease the concentration of different hormones responsible for the vaso-dilatation and the activation of the renin-angiotensine system that is seen in the early faze of the dumping syndrome. Somatostatin has also an effect on gastric motility and transit time.

One of the main problems is the high cost and daily subcutaneous administration of somatostatin analogues .

Somatuline® Autogel is a slow-release formulation that requires only monthly injection and supply high-dose, stable serum levels of lanreotide. These agents provide improved patient compliance since they are administered on a monthly schedule.

The purpose of this study is to assess if Somatuline autogel 90 mg is effective in the treatment of dumping syndrome. This will be a 27 weeks double blinded placebo-controlled cross-over multicenter study assessing the effect of Somatuline 90 mg in patients with dumping syndrome.

Reports on the therapeutic effectiveness of lanreotide in the management of dumping symptoms are scarce and based on small numbers of patients. Data on the effect of lanreotide in the treatment of dumping are missing. In this trial, all patients will be treated with Somatuline ® Autogel 90 mg. From a pharmacokinetic point of view, all patients will have reached steady state concentration of lanreotide after 12 weeks of treatment. After 12 weeks, a wash-out period of 4 weeks is inserted before patients will be crossed over to placebo or active treatment at week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical suspect of a dumping syndrome with a total dumping score* (early and late symptoms) ≥ 10, and

   1. a positive OGTT, in terms of a glycemia <60 mg/dl or Hematocrit increase > 3%, or an increase of pulse rate by 10 bpm Or
   2. documented spontaneous hypoglycemia (at least 1)
2. Age > 18 years
3. Diet of 6 meals a day with low concentration of mono- and disaccharides during 1 month before inclusion without sufficient improvement (= evaluation by physician and patient)

Exclusion Criteria:

1. Patients who have been treated with Somatuline or Sandostatine LAR in the past
2. Cholecystolithiasis
3. Diabetes Mellitus
4. Coeliakie and Giardia
5. Untreated severe oesophagitis
6. Untreated gastric and duodenum ulcer
7. Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to Study Day 1, and (d) female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
8. Hypersensitivity to lanreotide or one of the compounds of the drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Total Dumping score after treatment with Somatuline 90 mg and after placebo. | at week 11 and week 27 during the study
  Early dumping starts immediately after a meal, within 1 hour (< 1 hour). Late dumping starts later than 1 hour after a meal (≥ 1 hour). Each item is scored from zero (not present) 1 (mild) , 2 (moderate) and 3 (severe). Early dumping symptoms : sweating, flushes, dizziness, palpitations, abdominal pain, diarrhea, bloating, nausea. Late dumping symptoms : sweating, palpitations, hunger, drowsiness to unconsciousness, shaking and aggression.
  The change in dumping score will be assessed after 11 weeks and a second time after cross over at week 27.
  Additionally, the overall improvement is assessed by asking "how do you feel compared with your situation before starting the study at week 11. The same question is asked at week 27. Additionally at week 27 the following question is asked " How do you feel compared with your situation 4 months ago ?" Scoring is done on a 7 point Likert scale.

SECONDARY OUTCOMES:
Change in quality of life. | week 0, 11, 16 and 27
  To assess the effect of Somatuline 90 mg versus placebo on a standardized quality of life questionnaire (QOL SF-36).
The difference in number of participants with adverse events between somatuline 90 mg versus placebo | at week 27 (end of the study)
  To assess the tolerability of Somatuline 90 mg versus placebo.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - AZ St. Lucas, Brugges
  - ZOL Genk, Genk
  - University Hospitals Leuven, Leuven